CLINICAL TRIAL: NCT01901497
Title: Comparison of Pharmacokinetics of Amikacin Administered by Three Vibrating Mesh Nebulizers in Healthy Volunteers
Brief Title: Pharmacokinetics of Nebulized Amikacin in Non Invasive Ventilated Healthy Volunteers.
Acronym: NIV-NEBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital St Luc, Brussels (Other)
Collaborators: Haute Ecole de Santé Vaud (Other); Université Catholique de Louvain (Other); Ligue Pulmonaire Neuchâteloise (Other)
Responsible Party: Principal Investigator, Jean-Bernard Michotte, MSc, PhD Student, University Hospital St Luc, Brussels
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIVnebu
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Acute Respiratory Insufficiency; Chronic Respiratory Insufficiency; Bronchospasm and Obstruction
Keywords: non invasive ventilation; single limb circuit ventilator; bilevel; nebulization; nebulizer; vibrating mesh nebulizer; amikacin
MeSH Terms: conditions — Bronchial Spasm; Bites and Stings | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Solo nebulizer (Experimental): Amikacin (500 mg/4 mL) administered with an Aerogen AeroNeb Solo nebulizer associated with a bilevel ventilator
  Interventions: Device: Nebulizer
- Pro nebulizer (Experimental): Amikacin (500 mg/4 mL) administered with an Aerogen AeroNeb Pro nebulizer associated with a bilevel ventilator
  Interventions: Device: Nebulizer
- NIVO nebulizer (Experimental): Amikacin (500 mg/4 mL) administered with an Aerogen AeroNeb NIVO nebulizer associated with a bilevel ventilator
  Interventions: Device: Nebulizer

INTERVENTIONS:
Device: Nebulizer — 500 mg/4 mL Amikacin nebulized using vibrating mesh nebulizer associated with a single limb bilevel ventilator. The nebulizations are considered as finished when there is no visible evidence of nebulization for a period of 30 seconds.
  Other Names: Vibrating-mesh nebulizers

SUMMARY:
The purpose of the study is to compare the pharmacokinetics of nebulized amikacin administered with three vibrating mesh nebulizers coupled with a single limb circuit bilevel ventilator in healthy volunteers. Following our previous in vitro study, our hypotheses are that the pharmacokinetics varies among the devices tested and that a most efficient device can be identified.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication of amikacin
* Written informed consent
* Negative pregnant test (for women)

Exclusion Criteria:

* History of respiratory disease
* History of renal disease
* History of otological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of nebulized amikacin | within the first 24 hours after nebulization
  The area under the urinary amikacin concentration-time curve after nebulization(AUC0-24 hour) is calculated from the data obtained during 24 hours after nebulization. To determine amikacin absorption during the nebulization, amikacin concentrations are measured in the 24 hours urine collections, which reflected the quantity of dose absorbed via inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Michotte, PhD student, Principal Investigator — Cliniques Universitaires Saint-Luc (service de pneumologie), Haute Ecole de Santé Vaud (filière physiothérapie), Université Catholique de Louvain; Emilie Jossen, BSc, Principal Investigator — Ligue Pulmonaire Neuchâteloise; Jean Roeseler, PhD, Study Chair — Cliniques Universitaires Saint-Luc (service des soins intensifs); Giuseppe Liistro, MD, PhD, Study Chair — Université Catholique de Louvain, Institut de Recherche Expérimentale et Clinique (IREC), Pôle de Pneumologie, ORL & Dermatologie, 1200 Brussels, Belgium; Grégory Reychler, PhD, Study Director — Cliniques Universitaires Saint-Luc (service de pneumologie), Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc (Service des soins intensifs), Brussels, Belgium